CLINICAL TRIAL: NCT04865601
Title: Novel DNA Adductomics Methodological Developments for Research in Colon Cancer
Brief Title: DNA Adductomics for Colorectal Cancer Investigation
Acronym: adductomics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Professor Lars Ove Dragsted, professor, University of Copenhagen
Other Study IDs: M239
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer; Familial Adenomatous Polyposis; Hereditary Non-polyposis Colon Cancer; Lynch Syndrome
MeSH Terms: conditions — Colorectal Neoplasms; Adenomatous Polyposis Coli; Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Colon epithelium layer, white blood cells, serum, plasma, urine, faeces
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- CRC: Patient affected by any sporadic colorectal cancer
  Interventions: Other: resectomy of the colon
- FAP: Patients affected by familial adenomatous polyposis coli
  Interventions: Other: resectomy of the colon
- HNPCC: Patient affected by hereditary non polyposis colorectal cancer
  Interventions: Other: resectomy of the colon
- Lynch: patient affected by lynch syndrome
  Interventions: Other: resectomy of the colon
- others: Patients affected by ulcerative colitis, chron disease, diverticulitis and other colon diseases, which represent the control
  Interventions: Other: resectomy of the colon

INTERVENTIONS:
Other: resectomy of the colon — The patient scheduled for colon resectomy are included in the study

SUMMARY:
This project seeks to identify DNA-adducts in colon tissue from different groups of patients with CRC scheduled for complete or partial colon resections. Other patients scheduled for resection of the colon serve as controls. In addition, surrogate samples such as white blood cells are investigated for the presense of adducts while blood plasma and urine are investigated for the presense of DNA-repair products.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) develops as a result of multiple genetic mutations causing normal intestinal epithelium to transform into a colorectal carcinoma. Genetic mutations may be caused by many different genetic events including chemical damage to the DNA nucleosides. These chemical modifications are due to both exogenous compounds coming from diet, environment and gut microbiota, or endogenous compounds produced by our own metabolic processes like inflammation and oxidative stress. Such genetic alteration is thought to be the starting event leading to development of sporadic CRC. However, there is little understanding on which DNA nucleoside modifications are associated with increased risk of CRC and their mechanism of action. The study of these DNA nucleoside modifications has been addressed in the recent years by a new research field, called DNA adductomics. DNA adductomics uses the new advanced high resolution mass spectrometry (HRMS) instrumentations for identifying the complexes that are formed between toxic compounds and DNA, namely DNA adducts.

Some studies have been previously identified DNA adducts in CRC with older technology. However, there is not a real evidence on which DNA adducts are related to sporadic CRC, hereditary non polyposis colorectal cancer (HNPCC) and other diseases such as familial adenomatous polyposis (FAP) which turns into CRC with a 95% risk before the age of 35. The lack of more recent human studies in DNA adductomics is mainly due to the lack of appropriate analytical methods. Developing such methods requires sufficient sample material and the amount of sample in a colon biopsy is too low to be used for method development. In this study, colon epithelial tissue obtained by resection of colon during surgery will be used for developing a more sensitive method, possibly allowing DNA adduct analysis from biopsies in future studies. In order to ascertain that the developed method can differentiate the level of DNA-adducts between inherited CRC, sporadic CRC and non-CRC subjects, also materials from other groups coming to the hospital for colon resections will be obtained. By analyzing the materials obtained in a case-control manner, we might also be able to resolve whether some of the DNA adducts differ between the different CRC cases or in comparison with cancer-free subjects. This knowledge should provide a preliminary basis for suggesting prevention and intervention approaches to reduce morbidity and mortality from CRC.

However, in case-control studies, a proper selection of the subjects should be carried out by assuring gender and age balance between the control group and the CRC group. This will be difficult in the first part of the current study since 1) there is limited possibility of obtaining resected colon from healthy subjects 2) CRC incidence rates are markedly higher in men than in women, and 3) different types of CRC develop at different ages. It is also obvious that a method relying on analyses of colon resections would have a limited application in preventive medicine. A solution to these issues may be the use of appropriate surrogate samples like blood, faeces and urine. Indeed, since DNA lesions may be removed from the genome by the DNA repair system, they are often excreted in urine, in faeces, or in blood. In order to know whether we may substitute tissues with surrogate samples, we will explore whether there is a correlation between DNA-repair product level in surrogate samples and DNA adducts in colon tissues. Substituting colon tissues with surrogates, or developing a sensitive method for DNA analysis from biopsies, would allow an easier collection of the samples, giving the possibility, in the future, of performing large and controlled clinical studies as well as less invasive sampling from patients. This could allow to confirm a causal relationship between specific DNA-adducts and CRC, providing real advances in prevention and intervention approaches.

Finally, after the identification of the DNA adducts and DNA-repair products possibly associated with CRC, it will be important to identify the real cause of DNA adducts formation. Our final purpose is therefore identifying which life-style, dietary or environmental factors are possibly associated with the DNA adducts and DNA-repair products identified in colon and surrogate samples, respectively. For this purpose, we will perform a metabolic profiling of serum, urine and faeces, a microbial profiling of faeces, and we will correlate it with basic information on patient life styles about smoking, alcohol consumption and intake of red meat, e.g. factors suspected to influence risk of colonic diseases.

Establishing a causal relationship between specific DNA-adducts and CRC or other colonic diseases, and understanding the causes for DNA adducts formation, will not only yield much richer insights into the molecular defects but will also result in advances in prevention and intervention approaches.

ELIGIBILITY:
Inclusion Criteria:

* Patients with either FAP, Lynch syndrome, other HNPCC, sporadic colorectal cancer, ulcerative colitis or other conditions who are scheduled for whole or partial resection of their colon

Exclusion Criteria:

* Any condition that makes the investigator or hospital personnel doubt that voluntary participation isfeasible.
* Patients who are not able to understand and sign the informed consent form for any reason, including lack of a sufficient period of time to consider their participation.
* Patients who are below 18 years of age.
* Patients who donated blood to a blood bank within 3 months prior to their operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population will be selected among the patients with either FAP, Lynch syndrome, other HNPCC, sporadic colorectal cancer, ulcerative colitis or other conditions who are scheduled for whole or partial resection of their colon at Hvidovre hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
DNA adductome in CRC and other diseases | During surgery
  Identification of DNA adducts in colon tissue from CRC and other diseases
Correlation of DNA adduct and DNA repair products | Baseline (Before surgery)
  Correlation of DNA adduct in colon tissues and DNA repair products in surrogate samples

SECONDARY OUTCOMES:
Correlation of DNA adducts with microbiota | Baseline (Before surgery)
  Correlation of DNA adduct in colon tissues with microbiota and microbiota metabolites in faeces
Correlation of DNA adducts with CRC causes | Baseline (Before surgery)
  Correlation of DNA adduct in colon tissues with metabolism in serum and urine

CONTACTS AND LOCATIONS:
Overall Officials: Lars Ove O Dragsted, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Nutrition, Exercise and Sports, University of Copenhagen, Copenhagen, Frederiksberg C, Denmark

IPD SHARING:
Plan to Share IPD: Undecided